CLINICAL TRIAL: NCT05946109
Title: Tackling FRAILTY: ACTIVE-AGE@home: a Home-based Functional Exercise Program for Community Dwelling Frail Older Adults Provided by Professionals and Volunteers.
Brief Title: Effect of an Exercise Program for Frail Older Adults
Acronym: AA@HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University Ghent (Other); Universiteit Antwerpen (Other); Odisee University college for applied sciences (Other); Artevelde University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Patricia De Vriendt, Prof dr, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23075_AAathome
Record Dates: First submitted 2023-06-20; First posted 2023-07-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Frailty
Keywords: older adults; physical activity; exercise; rehabilitation; occupational therapy; health promotion; goal-oriented care; home based; primary care; geriatrics; activities of daily living; meaningful activities; cognition; loneliness; cost-effectiveness
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: This project aims to investigate the effect on physical functioning, cognition, loneliness, self-management, subjective health and meaningful activities of frail older adults, provided by professionals (study condition 1) or provided by trained volunteers (study condition 2) or when not provided (controls, study condition 3). Since it is hypothesized that volunteers will reduce health care cost, the investigators will assess health care utilization in the three groups. Therefore, a RCT will be used.. The duration of the intervention is 24 weeks and assessments will be done before, after and at 48 weeks follow-up. The trial is designed in line with The Geriatric ICF Core Set reflecting health-related problems in community-living older adults aged 75 years and older without dementia. To limit possible bias due to non-specific treatment effects, all participants allocated to both intervention arms will receive an identical amount of treatment, securing balanced treatment arms.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer algorithm will be used to generate the random allocation sequence. Participants will be randomized in a 1:1 ratio, using permuted block randomization into one of the three parallel groups. Randomization will be done centrally by an interactive web response system. Once the participants are found eligible for the trial, they can be randomized. This will generate a unique study randomization number and the treatment arm label (A professionals, B volunteers, C control) to which the participant is randomized. An accountability log with the corresponding label will be kept by the PI or delegated person to ensure that allocation was successfully performed. Participants will be scheduled to receive their randomisation within one week of eligibility assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ACTIVE-AGE@home by professionals (Active Comparator): Training program of 24 weeks supervised by professionals with a relevant background in the treatment and/or training of the older adults.
  The older adults are trained by either a physiotherapist, an occupational therapist or an exercise professional. The professionals will receive a 3x4h training course to gain more knowledge and practice regarding following aspects:
  * Frailty and ageing.
  * Physical training principles + ACTIVE-AGE@home exercise program
  * Motivational coaching.
  All participants in the three arms will receive the same monthly newsletter with tips and tricks to obtain good health in older age.
  Interventions: Behavioral: ACTIVE-AGE@home
- ACTIVE-AGE@home by volunteers (Experimental): Training program of 24 weeks supervised by volunteers who are presented by the older adults themselves or who are recruited by the research group.
  The older adults are trained by an informal caregiver or a newly recruited volunteer. The informal caregivers and volunteers will receive a 3x4h training course to gain more knowledge and practice regarding following aspects:
  * Frailty and ageing.
  * Physical training principles + ACTIVE-AGE@home exercise program
  * Motivational coaching.
  All participants in the three arms will receive the same monthly newsletter with tips and tricks to obtain good health in older age.
  Interventions: Behavioral: ACTIVE-AGE@home
- Standard care for frail older adults (No Intervention): The two intervention conditions will be compared with the current standard care for frail community-dwelling elderly that does not include physical activity interventions.
  All participants in the three arms will receive the same monthly newsletter with tips and tricks to obtain good health in older age.

INTERVENTIONS:
Behavioral: ACTIVE-AGE@home — functional, homebased training program offering basic functional exercises connected to meaningful activities, lifestyle coaching and motivational interviewing; derived from evidence-based training principles . Through a precise application of the FITT-VP* guidelines, a progressive and balanced program was designed and piloted in different proof-of-concept studies. The uniqueness of the program lies in the multi-component approach which brings together functional exercises for (1) muscle strength/muscle endurance, (2) aerobic endurance, (3) flexibility, motor ability and balance and (4) meaningful daily activities, in a home-based environment.
  The frail participants are visited three times a week during 24 weeks with in total 72 sessions. Each session is 1 hour in duration. Thus they receive 72 training hours.
  *(Frequency, Intensity, Time, Type of exercises, Volume and Progression)
  Other Names: ACTIEF@thuis
  Arms: ACTIVE-AGE@home by professionals; ACTIVE-AGE@home by volunteers

SUMMARY:
Despite the high level of evidence for physical activity as a countermeasure for frailty, the current Flemish standard of care does not include structural PA interventions for community-dwelling frail older adults. One barrier for this, is the high cost of supervised physical activity programmes.

Therefore, in this pragmatic randomised controlled trial, the investigators will consider the Flemish current standard of care for frail older adults as a control group. Intervention condition 1 reflects the state-of-the-art physical activity intervention provided by professionals and intervention condition 2 consists of the same intervention provided by trained volunteers. It is hypothesized that the intervention in both intervention conditions will have significant effects on functional ability, cognition, loneliness, self-management, subjective health and meaningful activities and that it can alleviate the financial burden of condition 1 (cost-effectiveness). The pretrajectory of this study was based on the 'British Medical Research Council guidance' for the development and evaluation of complex interventions. This resulted in a comprehensive, state-of-the art personalised physical activity programme for community-dwelling frail older adults: ACTIVE-AGE@home. The programme adheres to current guidelines for physical activity and exercise for frail older adults and considers low threshold and meaningful activities for the participants. The latter perfectly aligns with the complex bio-psychosocial components of frailty. Positive results will help reduce negative outcomes of frailty in older adults and will also reduce health and social expenditures. This study aligns with a 'prevention and health promotion' model.

DETAILED DESCRIPTION:
Studies show that physical activity can lower the risk of developing frailty and also reduce frailty-status once it is present. Favorable effects of physical activity on frail older adults include improved muscle strength, aerobic capacity, Quality of Life, cognition, and depression. There is also evidence of a dose response relationship between higher intensities of physical activity and lower levels of frailty. The current body of knowledge proves that physical activity interventions are the best possible (first-choice) treatment to tackle frailty. Despite of this, according to the World Health Organisation, only 7% of frail older adults meet the physical activity guidelines. In scientific literature and previously conducted own research several intrapersonal barriers were detected as a possible explanation for the low participation rates: fear, negative self-esteem, feeling useless, but also environmental barriers: lack of accessibility (location, information, …) and the absence of a familiar and trustworthy trainers, informal caregivers or volunteers to support the older adults and provide motivation and follow-up.

Rationale for study design:

This study is developed considering the United Nation's 'Decade of Healthy Ageing' and Europe's research agenda on prevention. Therefore, this project fits perfectly with initiatives such as 'Ageing in Place' and 'Societalisation of care'. This project also aligns with the overall framework of the vision on Healthy Ageing of the World Health Organisation (WHO).

Both physical activity and home-based services are reported as part of the top 10 priorities for frailty research by the Canadian Frailty Priority Setting and was co-created with frail older adults. More specifically, RCTs (followed by cost effectiveness studies) focusing on interventions for older adults with frailty are a high priority for the frailty research agenda. Strategies to slow the progression of frailty or convers the frailty state are paramount.

Volunteering:

Incorporating volunteering to provide physical activity interventions may reduce costs. In the 'Policy Framework for Active Ageing', the WHO advises to support peer leaders and groups that promote regular, moderate physical activity for people as they age and to inform and educate people and professionals about the importance of staying active as one grows older. The 'Flemish Council of the Elderly' together with the 'Flemish Institute for Health Promotion and Prevention' specifically recommends to train nonprofessional volunteers to counter frailty in lonely older adults. Also, Luger and coleaugues conducted a proof-of-concept study and showed that physical training, which is administered by trained lay nonprofessional volunteers, is feasible and can help to tackle frailty in older persons living at home. The fact that functional results of training can be obtained at a lower cost by the efforts of volunteers holds a cost saving potential which the investigators will be able to study. In Flanders 1 out of 8 people is volunteering and during the COVID-19 crisis the willingness to help others has risen.

Cost-effectiveness:

In Europe estimates are that in 2018, 11% of older adults (>65 years) were considered frail. Calculated for the whole EU-28 this means that a total of 56.364.000 older adults were frail. According to the 'Flemish Institute for Statistics' (the governing body where Flemish demographic data are collected and analyzed), the percentage of older adults in Flanders, aged 65 years or older, will increase from 20% or >1.300.000 older adults in 2017 to 23% or >1.500.000 older adults in 2027. Given the evidence based estimates that 35%-40% of older adults are in a reversible frail or pre-frail state, this means that the target population of this study has the magnitude of up to 600.000 Flemish older adults in 2027 that could benefit from ACTIVE-AGE@home. Regarding the societal and economic benefits, several studies pointed out that the average additional costs associated with frailty when controlled for ageing and multimorbidity range from 1.500 to 5.000 euro per person per year. As frailty is expected to be stabilized or reverted, a reduction in health care utilization by any intervention is realistic. The study by Sicsic demonstrated the impact of frailty transitions on health care utilisation. In their Europe-wide study, they found that becoming frail is associated with a 14.4 percentage point increase in hospital use, about 2 percentage points in GP consultations and 7.7 percentage point increase in specialist care. A delay or reverse of frailty clearly shows the cost saving potential of the intervention under study.

Study design:

The Proof of Concept Studies showed positive effects for the participants. Now, the research consortium will further evaluate ACTIVE-AGE@home for frail community-dwelling older adults, by testing its effect and evaluate also its cost-effectiveness when it is administered by professionals or by trained volunteers in combination with professionals and compare this to the care as usual in Flanders. A pragmatic RCT design is therefore the most relevant, effective, and efficient approach for this objective.

The duration of the intervention is 24 weeks and assessments will be done before (T=0), after (T=1) and at 48 weeks follow-up (T=2). To limit possible bias due to non-specific treatment effects, all participants allocated to the two intervention arms will receive an identical amount of treatment, securing balanced treatment arms. The third group will receive care as usual for frail older adults.

Condition 1: professionals The frail participants are visited three times a week by the trained professional, for 24 weeks with in total 72 sessions. Each session is 1 hour in duration. Thus, they receive 72 training hours equal to the volunteer-administered program. The professionals will receive three 4h training courses to gain more knowledge and practice regarding the specific innovative aspects of the programme, including information on frailty and ageing, motivational coaching, physical training principles and ACTIVE-AGE@home.

Condition 2: volunteers The frail participants are visited three times a week by trained non-professional volunteers, for 24 weeks with in total 72 sessions. Each session is 1 hour in duration. Thus, they receive 72 training hours, equal to the professional administered program. The volunteers will also receive three 4h training courses comparable to the professionals. Additionally, volunteers are coached by a professional during the intervention.

Condition 3: usual care / control Frail participants will receive no visits from volunteers or professionals and will not be trained with the ACTIVE-AGE@home exercise program. They can receive other care that is provided by health care professionals to frail older adults.

Health economic evaluations:

The health economic evaluations concern incremental analyses in terms of incremental costs over incremental effects between the alternatives. Therefore cost-utility analyses will be conducted. The thresholds suggested by the Belgian Health Care Knowledge Centre will be applied, and are based on the welfare of our country, expressed in GDP per capita (≈40,000€/QALY). This threshold represents a willingness-to-pay, as society, for one adjusted quality of life year gained. It creates however the illusion that there is a "hard" cut-off in determining interventions to be cost-effective or not. The latter calls for cautious interpretation of results as these cut-offs should be interpreted as indicative rather than a hard decision-rule. The investigators plan to conduct threshold analyses which look for a tipping point for one or more specific input parameters that lead to an incremental cost-effectiveness ratio above or below the threshold. Additionally, probabilistic sensitivity analyses will be conducted and presented in cost-effectiveness acceptability curves indicating at each possible threshold the likelihood whether one of the intervention arms is cost-effective compared to the alternative. This kind of analyses is informative to health decision policymakers in providing insight on factors that lead (or not) to a more cost-effective approach. These kinds of analyses will be presented to the advisory board for further discussion. Trial-based economic evaluation: first, the individual participant data from both groups will be used to estimate the health outcomes and costs of ACTIVE-AGE@home over the period from recruitment to 12 months. The cost-effectiveness analyses will be carried out from a societal perspective based on the Belgian guideline for health economic evaluations. The direct medical costs encompass all costs for treatment and follow-up from the health system perspective and all out-of-pocket contributions by the participant. National tariffs will be used for the valuation. Direct non-medical costs include transport costs, and home care help, whereas indirect costs include productivity loss due to informal care which will be documented and valued using the human capital approach and proxy good methods. The effects are expressed in utilities, derived from the national values of the MOS-SF-36. QALYs will be calculated using the area under the curve method. The cost-effectiveness of the intervention will be expressed in incremental cost per QALY gained (quality-adjusted life years). The incremental cost per QALY will be calculated as a ratio of (Expected Cost ACTIVE-AGE@home -Expected Cost standard care) / (Expected Outcome ACTIVEAGE@home - Expected Outcome standard care). The robustness of the results will be analyzed by probabilistic sensitivity analyses on the cost as well as on the outcome. Bootstrapping with replacement will be employed utilizing @Risk and MS Excel®, using a minimum of 1000 iterations to obtain 2.5% and 97.5% percentiles of the incremental cost-effectiveness ratio (ICER) distribution. All bootstrapped ICERs will be presented on a cost-effectiveness plane to determine the robustness of the ICER, and to determine the probability that ACTIVE-AGE@home is cost-effective at various willingness-to-pay thresholds. A cost-effectiveness acceptability curve will be used to depict the probabilities of acceptable ICERs.

Model based economic evaluation: In addition to the trial-based evaluation a model based evaluation will be performed which will allow us to account for the expected costs and health outcomes in both intervention and control groups beyond the follow-up period of the trial. A probabilistic Markov model will be developed compliant to the commonly used guidelines. The investigators assume a cycle of 1 year in the model and applying a lifetime horizon. Lifetime incremental costs and QALYs will be the input for the ICER calculation. Discount rates of 3% for costs and 1.5% for utilities will be applied, which is in line with the Belgian guidelines. Non-parametric bootstrapping will be applied for both costs and outcomes to test the robustness of the results. These iterations will be presented in cost-effectiveness planes. Probabilities to be cost effective for the different willingness-to-pay thresholds will be presented in cost-effectiveness acceptability curves.

ELIGIBILITY:
Inclusion Criteria:

* >70 years adults
* Frail according to the frailty phenotype of Fried, defining frailty as the presence of 3 or more of the following 5 criteria: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity

Exclusion Criteria:

life expectancy less than 12 months by any cause

* oncologic participants with active treatment
* treatment with exercise therapy in the preceding 6 months
* any contra-indication for exercise therapy as established by the treating physician/family practitioner
* cognitive impairment (unable to understand the test instructions and/or Mini Mental State Examination score <23/30)
* unable to understand the Dutch language
* diagnosed with Parkinson or Multiple Sclerosis
* having had a stroke in the preceding 6 months" to the registry

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The Timed Chair Stand (TCS) | T0 = 0 weeks, prior to start of exercise program
  The timed chair rise (TCS) is one of the most important functional evaluation clinical tests because it measures physical lower body strength and relates it to the most demanding ADLs (e.g., climbing stairs, getting out of a chair or bathtub, or rising from a horizontal position). This test is chosen based on literature data and consultancy of the experts of the research consortium. The TCR is considered a 'stress test', i.e., a test that aims to challenge the maximal physiological and/or physical capacity of the participant. It is responsive to change and influenceable via physical activity interventions, including ACTIVE-AGE@home. The test is also proven valid and reliable. In the TCR assessment, patients are asked to stand upright from a seated position in a chair (height 43 cm) with their arms folded across their chest and return to a seated position as many times as possible within a 30-s period.
The Timed Chair Stand (TCS) | T1 = 24 weeks, at the end of the exercise program
  The timed chair rise (TCS) is one of the most important functional evaluation clinical tests because it measures physical lower body strength and relates it to the most demanding ADLs (e.g., climbing stairs, getting out of a chair or bathtub, or rising from a horizontal position).
  This test is chosen based on literature data and consultancy of the experts of the research consortium. The TCR is considered a 'stress test', i.e., a test that aims to challenge the maximal physiological and/or physical capacity of the participant. It is responsive to change and influenceable via physical activity interventions, including ACTIVE-AGE@home. The test is also proven valid and reliable. In the TCR assessment, patients are asked to stand upright from a seated position in a chair (height 43 cm) with their arms folded across their chest and return to a seated position as many times as possible within a 30-s period.
The Timed Chair Stand (TCS) | T2 = 48 weeks, follow up measurement
  The timed chair rise (TCR) is one of the most important functional evaluation clinical tests because it measures physical lower body strength and relates it to the most demanding ADLs (e.g., climbing stairs, getting out of a chair or bathtub, or rising from a horizontal position). This test is chosen based on literature data and consultancy of the experts of the research consortium. The TCR is considered a 'stress test', i.e., a test that aims to challenge the maximal physiological and/or physical capacity of the participant. It is responsive to change and influenceable via physical activity interventions, including ACTIVE-AGE@home. The test is also proven valid and reliable. In the TCR assessment, patients are asked to stand upright from a seated position in a chair (height 43 cm) with their arms folded across their chest and return to a seated position as many times as possible within a 30-s period.

SECONDARY OUTCOMES:
Two Minute Step Test (TMST) | T0 = 0 weeks, prior to start of exercise program
  The Two Minute Step Test (TMST) designed to test the functional fitness of older adults, more specifically the aerobic endurance. The test is a valid and sensitive alternative to the 6 minute walk test. In the 2-Minute-Step-in-Place stress test the subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the kneecap and top of the hip bone. The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed and holding onto the wall, or a stable chair is allowed. The total number of times the right knee reaches the tape level in two minutes, is considered a proxy for aerobic endurance.
Two Minute Step Test (TMST) | T1 = 24 weeks, at the end of the exercise program
  The Two Minute Step Test (TMST)test is designed to test the functional fitness of older adults, more specifically the aerobic endurance. The test is a valid and sensitive alternative to the 6 minute walk test. In the 2-Minute-Step-in-Place stress test the subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the kneecap and top of the hip bone. The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed and holding onto the wall, or a stable chair is allowed. The total number of times the right knee reaches the tape level in two minutes, is considered a proxy for aerobic endurance.
Two Minute Step Test (TMST) | T2 = 48 weeks, follow up measurement
  The Two Minute Step Test (TMST) is designed to test the functional fitness of older adults, more specifically the aerobic endurance. The test is a valid and sensitive alternative to the 6 minute walk test. In the 2-Minute-Step-in-Place stress test the subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the kneecap and top of the hip bone. The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Resting is allowed and holding onto the wall, or a stable chair is allowed. The total number of times the right knee reaches the tape level in two minutes, is considered a proxy for aerobic endurance.
The Timed Up and Go Test | T0 = 0 weeks, prior to start of exercise program
  The purpose of the Timed Up and Go Test is to assess agility/dynamic balance, which is important in tasks that require quick displacement such as getting on and off public transport or getting up to attend to daily activities or chores in the kitchen, the bathroom or to answer the phone. The Timed Up and Go test is measured by the number of seconds the participant needs to get up from a seated position, walk 8 feet (2.44 m), turn, and return to the seated position.
The Timed Up and Go Test | T1 = 24 weeks, at the end of the exercise program
  The purpose of the Timed Up and Go Test is to assess agility/dynamic balance, which is important in tasks that require quick displacement such as getting on and off public transport or getting up to attend to daily activities or chores in the kitchen, the bathroom or to answer the phone. The Timed Up and Go test is measured by the number of seconds the participant needs to get up from a seated position, walk 8 feet (2.44 m), turn, and return to the seated position.
The Timed Up and Go Test | T2 = 48 weeks, follow up measurement
  The purpose of the Timed Up and Go Test is to assess agility/dynamic balance, which is important in tasks that require quick displacement such as getting on and off public transport or getting up to attend to daily activities or chores in the kitchen, the bathroom or to answer the phone. The Timed Up and Go test is measured by the number of seconds the participant needs to get up from a seated position, walk 8 feet (2.44 m), turn, and return to the seated position.
MOS 36-item-short-form health survey (SF-36) | T0 = 0 weeks, prior to start of exercise program
  Health related Quality of Life will be measured by using the MOS 36-item-short-form health survey (SF-36)56 , one of the most commonly used measures of HRQoL in the older population. The SF-36 questionnaire is widely used to monitor general population health status, to evaluate the efficacy of interventions, to monitor health status in patients with chronic disease and to determine the relative burdens of various diseases. Based on our POC study, we expect the following domains to be effective: (1) physical functioning, (2) physical role functioning, (3) bodily pain, (4) mental health and (5) vitality.
MOS 36-item-short-form health survey (SF-36) | T1 = 24 weeks, at the end of the exercise program
  Health related Quality of Life will be measured by using the MOS 36-item-short-form health survey (SF-36)56 , one of the most commonly used measures of HRQoL in the older population. The SF-36 questionnaire is widely used to monitor general population health status, to evaluate the efficacy of interventions, to monitor health status in patients with chronic disease and to determine the relative burdens of various diseases. Based on our POC study, we expect the following domains to be effective: (1) physical functioning, (2) physical role functioning, (3) bodily pain, (4) mental health and (5) vitality.
MOS 36-item-short-form health survey (SF-36) | T2 = 48 weeks, follow up measurement
  Health related Quality of Life will be measured by using the MOS 36-item-short-form health survey (SF-36)56 , one of the most commonly used measures of HRQoL in the older population. The SF-36 questionnaire is widely used to monitor general population health status, to evaluate the efficacy of interventions, to monitor health status in patients with chronic disease and to determine the relative burdens of various diseases. Based on our POC study, we expect the following domains to be effective: (1) physical functioning, (2) physical role functioning, (3) bodily pain, (4) mental health and (5) vitality.
iMTA Medical Consumption Questionnaire (iMCQ) | T0 = 0 weeks, prior to start of exercise program
  Medical consumption of frail older participants will be measured by the iMTA Medical Consumption Questionnaire (iMCQ). This questionnaire includes questions related to frequent contacts with healthcare providers. Because of comorbidities and frequent healthcare visits it is not always possible for the patient to define healthcare consumption according to his/her specific illness or condition. Therefore the iMCQ is a rather generic questionnaire.
iMTA Medical Consumption Questionnaire (iMCQ) | T1 = 24 weeks, at the end of the exercise program
  Medical consumption of frail older participants will be measured by the iMTA Medical Consumption Questionnaire (iMCQ). This questionnaire includes questions related to frequent contacts with healthcare providers. Because of comorbidities and frequent healthcare visits it is not always possible for the patient to define healthcare consumption according to his/her specific illness or condition. Therefore the iMCQ is a rather generic questionnaire.
iMTA Medical Consumption Questionnaire (iMCQ) | T2 = 48 weeks, follow up measurement
  Medical consumption of frail older participants will be measured by the iMTA Medical Consumption Questionnaire (iMCQ). This questionnaire includes questions related to frequent contacts with healthcare providers. Because of comorbidities and frequent healthcare visits it is not always possible for the patient to define healthcare consumption according to his/her specific illness or condition. Therefore the iMCQ is a rather generic questionnaire.
MOCA Montreal Cognitive Assessment | T0 = 0 weeks, prior to start of exercise program
  The Montreal Cognitive Assessment (MoCA) was developed as a tool for screening patients who present with mild cognitive complaints but who usually perform within the normal range on the MMSE. However, we will not use this test as a screening tool, but as a way to evaluate the effect of the intervention on cognitive functions. The total score for the MoCA ranges from 0 to 30 points distributed among the following domains: memory, naming, language, visuospatial/executive functions, abstraction, attention/concentration/calculation and orientation. The MoCA is a time-effective test comprising 22 items. Psychometric indexes revealed that the MoCA is a reliable and valid instrument. A reliable change of ±1.73 points in a time period of 3.5 years represented a clinically meaningful difference. This threshold increases the likelihood that an individual's change in performance reflects actual change in cognitive ability rather than related to extraneous factors.
MOCA Montreal Cognitive Assessment | T1 = 24 weeks, at the end of the exercise program
  The Montreal Cognitive Assessment (MoCA) was developed as a tool for screening patients who present with mild cognitive complaints but who usually perform within the normal range on the MMSE. However, we will not use this test as a screening tool, but as a way to evaluate the effect of the intervention on cognitive functions. The total score for the MoCA ranges from 0 to 30 points distributed among the following domains: memory, naming, language, visuospatial/executive functions, abstraction, attention/concentration/calculation and orientation. The MoCA is a time-effective test comprising 22 items. Psychometric indexes revealed that the MoCA is a reliable and valid instrument. A reliable change of ±1.73 points in a time period of 3.5 years represented a clinically meaningful difference. This threshold increases the likelihood that an individual's change in performance reflects actual change in cognitive ability rather than related to extraneous factors.
MOCA Montreal Cognitive Assessment | T2 = 48 weeks, follow up measurement
  The Montreal Cognitive Assessment (MoCA) was developed as a tool for screening patients who present with mild cognitive complaints but who usually perform within the normal range on the MMSE. However, we will not use this test as a screening tool, but as a way to evaluate the effect of the intervention on cognitive functions. The total score for the MoCA ranges from 0 to 30 points distributed among the following domains: memory, naming, language, visuospatial/executive functions, abstraction, attention/concentration/calculation and orientation. The MoCA is a time-effective test comprising 22 items. Psychometric indexes revealed that the MoCA is a reliable and valid instrument. A reliable change of ±1.73 points in a time period of 3.5 years represented a clinically meaningful difference. This threshold increases the likelihood that an individual's change in performance reflects actual change in cognitive ability rather than related to extraneous factors.
Trail making test | T0 = 0 weeks, prior to start of exercise program
  The Trail Making Test (TMT) is widely used as a cognitive task to measure attention and executive function among older adults. It involves connecting randomly arranged circles with a pencil, and comes in Parts A (TMT-A) and B (TMT-B). In TMT-A, numbers are written in circles, and test takers are asked to connect the numbers in ascending order. In TMT-B, numbers or letters are written in circles, and test takers are asked to connect them alternately and in ascending order. In both TMTs, the time to completion is the main evaluation index. Processing speed such as that required for visual search is strongly reflected in the results of TMT-A, and working memory and cognitive flexibility are involved in TMT-B.
Trail making test | T1 = 24 weeks, at the end of the exercise program
  The Trail Making Test (TMT) is widely used as a cognitive task to measure attention and executive function among older adults. It involves connecting randomly arranged circles with a pencil, and comes in Parts A (TMT-A) and B (TMT-B). In TMT-A, numbers are written in circles, and test takers are asked to connect the numbers in ascending order. In TMT-B, numbers or letters are written in circles, and test takers are asked to connect them alternately and in ascending order. In both TMTs, the time to completion is the main evaluation index. Processing speed such as that required for visual search is strongly reflected in the results of TMT-A, and working memory and cognitive flexibility are involved in TMT-B.
Trail making test | T2 = 48 weeks, follow up measurement
  The Trail Making Test (TMT) is widely used as a cognitive task to measure attention and executive function among older adults. It involves connecting randomly arranged circles with a pencil, and comes in Parts A (TMT-A) and B (TMT-B). In TMT-A, numbers are written in circles, and test takers are asked to connect the numbers in ascending order. In TMT-B, numbers or letters are written in circles, and test takers are asked to connect them alternately and in ascending order. In both TMTs, the time to completion is the main evaluation index. Processing speed such as that required for visual search is strongly reflected in the results of TMT-A, and working memory and cognitive flexibility are involved in TMT-B.
Rey Auditory Verbal Learning Test | T0 = 0 weeks, prior to start of exercise program
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological assessment designed to evaluate verbal memory. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time. The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. After five repetitions of free-recall, a second "interference" list (List B) is presented in the same manner, and the participant is asked to recall as many words from List B as possible. After the interference trial, the participant is immediately asked to recall the words from List A, which she or he heard five times previously. After a 20 min delay, the participant is asked to again recall the words from List A.
Rey Auditory Verbal Learning Test | T1 = 24 weeks, at the end of the exercise program
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological assessment designed to evaluate verbal memory. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time. The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. After five repetitions of free-recall, a second "interference" list (List B) is presented in the same manner, and the participant is asked to recall as many words from List B as possible. After the interference trial, the participant is immediately asked to recall the words from List A, which she or he heard five times previously. After a 20 min delay, the participant is asked to again recall the words from List A.
Rey Auditory Verbal Learning Test | T2 = 48 weeks, follow up measurement
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological assessment designed to evaluate verbal memory. The RAVLT can be used to evaluate the nature and severity of memory dysfunction and to track changes in memory function over time. The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. After five repetitions of free-recall, a second "interference" list (List B) is presented in the same manner, and the participant is asked to recall as many words from List B as possible. After the interference trial, the participant is immediately asked to recall the words from List A, which she or he heard five times previously. After a 20 min delay, the participant is asked to again recall the words from List A.
De Jong Gierveld 11-item loneliness scale | T0 = 0 weeks, prior to start of exercise program
  This scale consists of 11 items that examine the feelings of loneliness and distinguishes between social and emotional loneliness. Of the 11 items, six items measure emotional loneliness with negative semantic load, and five items identify social loneliness with sentences using positive semantic load.
  The 11-item De Jong Gierveld scale has proved to be a valid and reliable measuring instrument for overall, emotional and social loneliness. Its reliability was found to be adequate (Cronbach's α = 0.87) and also showed convergent validity with measures of depressive symptoms and social support, suggesting that the construct measured by this test is appropriate to be used as an indicator of loneliness.
De Jong Gierveld 11-item loneliness scale | T1 = 24 weeks, at the end of the exercise program
  This scale consists of 11 items that examine the feelings of loneliness and distinguishes between social and emotional loneliness. Of the 11 items, six items measure emotional loneliness with negative semantic load, and five items identify social loneliness with sentences using positive semantic load.
  The 11-item De Jong Gierveld scale has proved to be a valid and reliable measuring instrument for overall, emotional and social loneliness. Its reliability was found to be adequate (Cronbach's α = 0.87) and also showed convergent validity with measures of depressive symptoms and social support, suggesting that the construct measured by this test is appropriate to be used as an indicator of loneliness.
De Jong Gierveld 11-item loneliness scale | T2 = 48 weeks, follow up measurement
  This scale consists of 11 items that examine the feelings of loneliness and distinguishes between social and emotional loneliness. Of the 11 items, six items measure emotional loneliness with negative semantic load, and five items identify social loneliness with sentences using positive semantic load.
  The 11-item De Jong Gierveld scale has proved to be a valid and reliable measuring instrument for overall, emotional and social loneliness. Its reliability was found to be adequate (Cronbach's α = 0.87) and also showed convergent validity with measures of depressive symptoms and social support, suggesting that the construct measured by this test is appropriate to be used as an indicator of loneliness.
Engagement in meaningful activities scale | T0 = 0 weeks, prior to start of exercise program
  The Engagement In meaningful activities scale (EMAS) is a 12-item questionnaire with statements about activities and meaning in these activities. The highest score is 48, participants are considered to have low meaning when they score lower than 29, moderate meaning when they score between, they score between 29 - 41 and when they score higher than 41, a high meaning.Psychometric properties: internal consistency of the EMAS was very good, (α = .89). Two week test-retest reliability for the EMAS was moderate [r(24) = .56, p < . 01]. Corrected item-total correlations for the EMAS ranged from .48 to .72
Engagement in meaningful activities scale | T1 = 24 weeks, at the end of the exercise program
  The Engagement In meaningful activities scale (EMAS) is a 12-item questionnaire with statements about activities and meaning in these activities. The highest score is 48, participants are considered to have low meaning when they score lower than 29, moderate meaning when they score between, they score between 29 - 41 and when they score higher than 41, a high meaning. Psychometric properties: internal consistency of the EMAS was very good, (α = .89). Two week test-retest reliability for the EMAS was moderate [r(24) = .56, p < . 01]. Corrected item-total correlations for the EMAS ranged from .48 to .72
Engagement in meaningful activities scale | T2 = 48 weeks, follow up measurement
  The Engagement In meaningful activities scale (EMAS) is a 12-item questionnaire with statements about activities and meaning in these activities. The highest score is 48, participants are considered to have low meaning when they score lower than 29, moderate meaning when they score between, they score between 29 - 41 and when they score higher than 41, a high meaning.
  Psychometric properties: internal consistency of the EMAS was very good, (α = .89). Two week test-retest reliability for the EMAS was moderate [r(24) = .56, p < . 01]. Corrected item-total correlations for the EMAS ranged from .48 to .72
Self-Management Abilities Scale - Short Form2 | T0 = 0 weeks, prior to start of exercise program
  The Self-management abilities scale short form (SMAS-S) is a questionnaire designed to measure six self-management abilities in older adults based on five dimensions of well-being specified in the social productions function (SPF) theory. These consist of the ability to ensure multifunctionality, maintain variety in resources, keep a positive frame of mind, invest in resources for longer term benefits, self-efficacy and taking initiative. SMAS-S is a shorter version from the originally developed SMAS-30 and consists of 18 items. Having a shorter instrument makes it more feasible to assess self-management abilities in a broader number of people, especially among frail older adults.
Self-Management Abilities Scale - Short Form2 | T1 = 24 weeks, at the end of the exercise program
  The Self-management abilities scale short form (SMAS-S) is a questionnaire designed to measure six self-management abilities in older adults based on five dimensions of well-being specified in the social productions function (SPF) theory. These consist of the ability to ensure multifunctionality, maintain variety in resources, keep a positive frame of mind, invest in resources for longer term benefits, self-efficacy and taking initiative. SMAS-S is a shorter version from the originally developed SMAS-30 and consists of 18 items. Having a shorter instrument makes it more feasible to assess self-management abilities in a broader number of people, especially among frail older adults.
Self-Management Abilities Scale - Short Form2 | T2 = 48 weeks, follow up measurement
  The Self-management abilities scale short form (SMAS-S) is a questionnaire designed to measure six self-management abilities in older adults based on five dimensions of well-being specified in the social productions function (SPF) theory. These consist of the ability to ensure multifunctionality, maintain variety in resources, keep a positive frame of mind, invest in resources for longer term benefits, self-efficacy and taking initiative. SMAS-S is a shorter version from the originally developed SMAS-30 and consists of 18 items. Having a shorter instrument makes it more feasible to assess self-management abilities in a broader number of people, especially among frail older adults.
Fatigue resistance grip strength test | T0 = 0 weeks, prior to start of exercise program
  In the Fatigue resistance grip strength, the Martin Vigorimeter is used to measure muscle fatigability. The subject is seated with both feet on the ground, the shoulder in neutral position and the elbow flexed in 90°. The participant holds the large bulb of the Martin Vigorimeter in the dominant hand by enclosing it on one side with the thumb and on the other side with four fingers. The participant is instructed to push the large pear as hard as possible and to maintain this force as long as possible. A good to excellent inter- and intra-observer reliability is observed (ICC values ranging from 0.77 to 0.94). Hand grip strength is seen as an indicator of overall body strength for frail older adults and other populations. Lower body strength leads to adverse health outcomes e.g. falls, disability and a higher risk of frailty.
Fatigue resistance grip strength test | T1 = 24 weeks, at the end of the exercise program
  In the Fatigue resistance grip strength, the Martin Vigorimeter is used to measure muscle fatigability. The subject is seated with both feet on the ground, the shoulder in neutral position and the elbow flexed in 90°. The participant holds the large bulb of the Martin Vigorimeter in the dominant hand by enclosing it on one side with the thumb and on the other side with four fingers. The participant is instructed to push the large pear as hard as possible and to maintain this force as long as possible. A good to excellent inter- and intra-observer reliability is observed (ICC values ranging from 0.77 to 0.94). Hand grip strength is seen as an indicator of overall body strength for frail older adults and other populations. Lower body strength leads to adverse health outcomes e.g. falls, disability and a higher risk of frailty.
Fatigue resistance grip strength test | T2 = 48 weeks, follow up measurement
  In the Fatigue resistance grip strength, the Martin Vigorimeter is used to measure muscle fatigability. The subject is seated with both feet on the ground, the shoulder in neutral position and the elbow flexed in 90°. The participant holds the large bulb of the Martin Vigorimeter in the dominant hand by enclosing it on one side with the thumb and on the other side with four fingers. The participant is instructed to push the large pear as hard as possible and to maintain this force as long as possible. A good to excellent inter- and intra-observer reliability is observed (ICC values ranging from 0.77 to 0.94). Hand grip strength is seen as an indicator of overall body strength for frail older adults and other populations. Lower body strength leads to adverse health outcomes e.g. falls, disability and a higher risk of frailty.
Activities of Daily Life (National Health Interview Survey) (HIS) | T0 = 0 weeks, prior to start of exercise program
  Every five years a national Health Interview Survey (HIS) is held in Belgium. This cross-sectional population survey includes questions on health status, lifestyle, use of health services and socio-demographic characteristics and is administered in a representative sample of the Belgian population. In the ACTIVE-AGE@home study, questions regarding Activities of Daily Living (ADL) are adopted from the HIS.
  The respondent is asked to indicate if they have difficulties performing daily activities and/or household tasks. The 7 daily activities and 7 household tasks are read out loud, answers are given by selecting a predefined 4-point scale ranging from 'no, no difficulties', 'yes, a few difficulties', 'yes, a lot of difficulties' of 'not possible to perform'. When a question is not applicable 'does not apply' can be noted as well.
  Activities of Daily Living are getting in and out of bed, sitting down or standing up from a chair, getting (un)dressed, taking a bath or shower, washing
Activities of Daily Life (National Health Interview Survey) (HIS) | T1 = 24 weeks, at the end of the exercise program
  Every five years a national Health Interview Survey (HIS) is held in Belgium. This cross-sectional population survey includes questions on health status, lifestyle, use of health services and socio-demographic characteristics and is administered in a representative sample of the Belgian population. In the ACTIVE-AGE@home study, questions regarding Activities of Daily Living (ADL) are adopted from the HIS.
  The respondent is asked to indicate if they have difficulties performing daily activities and/or household tasks. The 7 daily activities and 7 household tasks are read out loud, answers are given by selecting a predefined 4-point scale ranging from 'no, no difficulties', 'yes, a few difficulties', 'yes, a lot of difficulties' of 'not possible to perform'. When a question is not applicable 'does not apply' can be noted as well.
  Activities of Daily Living are getting in and out of bed, sitting down or standing up from a chair, getting (un)dressed, taking a bath or shower, washing
Activities of Daily Life (National Health Interview Survey) (HIS) | T2 = 48 weeks, follow up measurement
  Every five years a national Health Interview Survey (HIS) is held in Belgium. This cross-sectional population survey includes questions on health status, lifestyle, use of health services and socio-demographic characteristics and is administered in a representative sample of the Belgian population. In the ACTIVE-AGE@home study, questions regarding Activities of Daily Living (ADL) are adopted from the HIS.
  The respondent is asked to indicate if they have difficulties performing daily activities and/or household tasks. The 7 daily activities and 7 household tasks are read out loud, answers are given by selecting a predefined 4-point scale ranging from 'no, no difficulties', 'yes, a few difficulties', 'yes, a lot of difficulties' of 'not possible to perform'. When a question is not applicable 'does not apply' can be noted as well.
  Activities of Daily Living are getting in and out of bed, sitting down or standing up from a chair, getting (un)dressed, taking a bath or shower, washing

CONTACTS AND LOCATIONS:
Overall Officials: Patricia De Vriendt, Prof dr, Principal Investigator — VUB
Locations (1):
- UZ Brussels, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehler DS, Theou O. The impact of physical activity and sedentary behaviors on frailty levels. Mech Ageing Dev. 2019 Jun;180:29-41. doi: 10.1016/j.mad.2019.03.004. Epub 2019 Mar 26. PMID 30926562
- [Background] Negm AM, Kennedy CC, Thabane L, Veroniki AA, Adachi JD, Richardson J, Cameron ID, Giangregorio A, Petropoulou M, Alsaad SM, Alzahrani J, Maaz M, Ahmed MM, Kim E, Tehfe H, Dima R, Sabanayagam K, Hewston P, Abu Alrob H, Papaioannou A. Management of Frailty: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2019 Oct;20(10):1190-1198. doi: 10.1016/j.jamda.2019.08.009. PMID 31564464
- [Background] Rogers NT, Marshall A, Roberts CH, Demakakos P, Steptoe A, Scholes S. Physical activity and trajectories of frailty among older adults: Evidence from the English Longitudinal Study of Ageing. PLoS One. 2017 Feb 2;12(2):e0170878. doi: 10.1371/journal.pone.0170878. eCollection 2017. PMID 28152084
- [Background] Dent E, Hoogendijk EO, Visvanathan R, Wright ORL. Malnutrition Screening and Assessment in Hospitalised Older People: a Review. J Nutr Health Aging. 2019;23(5):431-441. doi: 10.1007/s12603-019-1176-z. PMID 31021360
- [Background] Luger E, Dorner TE, Haider S, Kapan A, Lackinger C, Schindler K. Effects of a Home-Based and Volunteer-Administered Physical Training, Nutritional, and Social Support Program on Malnutrition and Frailty in Older Persons: A Randomized Controlled Trial. J Am Med Dir Assoc. 2016 Jul 1;17(7):671.e9-671.e16. doi: 10.1016/j.jamda.2016.04.018. PMID 27346650
- [Background] Sicsic J, Rapp T. Frailty transitions and health care use in Europe. Health Serv Res. 2019 Dec;54(6):1305-1315. doi: 10.1111/1475-6773.13208. Epub 2019 Sep 30. PMID 31571222
- [Background] Mijnarends DM, Meijers JM, Halfens RJ, ter Borg S, Luiking YC, Verlaan S, Schoberer D, Cruz Jentoft AJ, van Loon LJ, Schols JM. Validity and reliability of tools to measure muscle mass, strength, and physical performance in community-dwelling older people: a systematic review. J Am Med Dir Assoc. 2013 Mar;14(3):170-8. doi: 10.1016/j.jamda.2012.10.009. Epub 2012 Dec 29. PMID 23276432
- [Background] Bohannon RW, Crouch R. 1-Minute Sit-to-Stand Test: SYSTEMATIC REVIEW OF PROCEDURES, PERFORMANCE, AND CLINIMETRIC PROPERTIES. J Cardiopulm Rehabil Prev. 2019 Jan;39(1):2-8. doi: 10.1097/HCR.0000000000000336. PMID 30489442
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Singleton N, Turner A. Measuring patients' views of their health. SF 36 is suitable for elderly patients. BMJ. 1993 Jul 10;307(6896):126-7. doi: 10.1136/bmj.307.6896.126-b. No abstract available. PMID 8123095
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Schoenberg MR, Dawson KA, Duff K, Patton D, Scott JG, Adams RL. Test performance and classification statistics for the Rey Auditory Verbal Learning Test in selected clinical samples. Arch Clin Neuropsychol. 2006 Oct;21(7):693-703. doi: 10.1016/j.acn.2006.06.010. Epub 2006 Sep 20. PMID 16987634
- [Background] De Jong Gierveld J, Van Tilburg T. The De Jong Gierveld short scales for emotional and social loneliness: tested on data from 7 countries in the UN generations and gender surveys. Eur J Ageing. 2010 Jun;7(2):121-130. doi: 10.1007/s10433-010-0144-6. Epub 2010 Apr 9. PMID 20730083
- [Background] Eakman AM. Measurement characteristics of the engagement in meaningful activities survey in an age-diverse sample. Am J Occup Ther. 2012 Mar-Apr;66(2):e20-9. doi: 10.5014/ajot.2012.001867. PMID 22394537
- [Background] Schuurmans H, Steverink N, Frieswijk N, Buunk BP, Slaets JP, Lindenberg S. How to measure self-management abilities in older people by self-report. The development of the SMAS-30. Qual Life Res. 2005 Dec;14(10):2215-28. doi: 10.1007/s11136-005-8166-9. PMID 16328901
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Derived] Vrancken D, De Smedt E, Tambeur J, De Keyser E, Vanbeuren E, Beckwee D, Lieten S, Annemans L, Peersman W, Van de Velde D, De Vriendt P. Effectiveness and cost-effectiveness of a home-based functional exercise programme for community-dwelling frail older adults, ACTIVE-AGE@home, provided by professionals and volunteers: protocol of a pragmatic randomised controlled trial. BMJ Open. 2025 Apr 7;15(4):e090746. doi: 10.1136/bmjopen-2024-090746. PMID 40194869
- See also: Partner institution Artevelde University of Applied Sciences has a project page where elaborate information and tools regarding the study are available and will be posted in the future. — https://www.arteveldehogeschool.be/nl/onderzoek/projecten/effectiviteit-trainingsprogramma-active-agehome-voor-kwetsbare-thuiswonende
- See also: Host institution VUB has a project page where basic information on the study is available. — https://www.vubtechtransfer.be/active-agehome-a-home-based-functional-exercise-program-for-community-dwelling-frail-older-adults